CLINICAL TRIAL: NCT01502371
Title: A 12-Week, Randomized, Placebo-Controlled, Dose-Ranging, Efficacy and Safety Study of Mometasone Furoate Metered Dose Inhaler in the Treatment of Children Ages 5 to 11 Years With Persistent Asthma (Phase 2; Protocol No. P04223AM3)
Brief Title: A Study of Mometasone Furoate Metered Dose Inhaler in Children With Persistent Asthma (P04223)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04223; 2008-007504-28 (EudraCT Number); MK-0887-086 (Other: Merck)
Record Dates: First submitted 2011-12-28; First posted 2011-12-30 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2022-02

CONDITIONS: Asthma
Keywords: Asthma; Children; Persistent
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Metered Dose Inhalers; Dry Powder Inhalers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- MF MDI 50 mcg BID (Experimental): Participants receive MF MDI 25 mcg x 2 inhalations (50 mcg total dose) BID PLUS Placebo dry powder inhaler (DPI) x 1 inhalation once daily (QD) in the evening for 12 weeks.
  Interventions: Drug: Mometasone Furoate (MF) Metered Dose Inhaler (MDI), 25 mcg; Drug: Placebo Dry Powder Inhaler (DPI)
- MF MDI 100 mcg BID (Experimental): Participants receive MF MDI 50 mcg x 2 inhalations (100 mcg total dose) BID PLUS Placebo DPI x 1 inhalation QD in the evening for 12 weeks.
  Interventions: Drug: Mometasone Furoate (MF) Metered Dose Inhaler (MDI), 50 mcg; Drug: Placebo Dry Powder Inhaler (DPI)
- MF MDI 200 mcg BID (Experimental): Participants receive MF MDI 100 mcg x 2 inhalations (200 mcg total dose) BID PLUS Placebo DPI x 1 inhalation QD in the evening for 12 weeks.
  Interventions: Drug: Mometasone Furoate (MF) Metered Dose Inhaler (MDI), 100 mcg; Drug: Placebo Dry Powder Inhaler (DPI)
- MF DPI 100 mcg QD (Active Comparator): Participants receive Placebo MDI x 2 inhalations BID PLUS MF DPI x 1 inhalation QD in the evening for 12 weeks.
  Interventions: Drug: Mometasone Furoate (MF) Dry Powder Inhaler (DPI), 100 mcg; Drug: Placebo Metered Dose Inhaler (MDI)
- Placebo (Placebo Comparator): Participants receive Placebo MDI x 2 inhalations BID PLUS Placebo DPI x 1 inhalation QD in the evening for 12 weeks.
  Interventions: Drug: Placebo Metered Dose Inhaler (MDI); Drug: Placebo Dry Powder Inhaler (DPI)

INTERVENTIONS:
Drug: Mometasone Furoate (MF) Metered Dose Inhaler (MDI), 25 mcg — MF MDI 25 mcg (per inhalation), 2 puffs BID for 12 weeks
  Arms: MF MDI 50 mcg BID
Drug: Mometasone Furoate (MF) Metered Dose Inhaler (MDI), 50 mcg — MF MDI 50 mcg (per inhalation), 2 puffs BID for 12 weeks
  Arms: MF MDI 100 mcg BID
Drug: Mometasone Furoate (MF) Metered Dose Inhaler (MDI), 100 mcg — MF MDI 100 mcg (per inhalation), 2 puffs BID for 12 weeks
  Arms: MF MDI 200 mcg BID
Drug: Mometasone Furoate (MF) Dry Powder Inhaler (DPI), 100 mcg — MF DPI 100 mcg (per inhalation), 1 puff QD for 12 weeks
  Other Names: Asmanex® Twisthaler®
  Arms: MF DPI 100 mcg QD
Drug: Placebo Metered Dose Inhaler (MDI) — Placebo MDI, 2 puffs BID for 12 weeks
  Arms: MF DPI 100 mcg QD; Placebo
Drug: Placebo Dry Powder Inhaler (DPI) — Placebo DPI, 1 puff QD for 12 weeks
  Arms: MF MDI 100 mcg BID; MF MDI 200 mcg BID; MF MDI 50 mcg BID; Placebo

SUMMARY:
The primary objective of this study is to demonstrate the dose-related efficacy, by evaluating morning (AM) lung function at the end of the dosing interval (AM pre-dose percent predicted forced expiratory volume in one second [FEV1]) across 12 weeks of treatment, of three doses (50 mcg, 100 mcg, and 200 mcg) of Mometasone Furoate (MF) Metered Dose Inhaler (MDI) twice a day (BID) compared with Placebo in children 5 to 11 years of age, inclusive, with persistent asthma. The primary hypothesis of this study is that at least one dose of MF MDI BID increases lung function, defined as a significant increase in percent predicted FEV1, when compared to Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma of at least 6 months duration.
* Using an Inhaled corticosteroid (ICS), either alone or in combination with a long-acting beta-2 agonist (LABA), for at least 12 weeks prior to the Screening Visit and must have been on a stable asthma regimen for at least 2 weeks prior to the Screening Visit, must not have used oral glucocorticosteroids within 30 days of the Screening Visit.

Exclusion Criteria:

* Treated in the emergency room for a severe asthma exacerbation requiring systemic glucocorticosteroid treatment, or hospitalization for management of airway obstruction within 3 months prior to the Screening Visit.
* History of ventilator support for respiratory failure secondary to asthma.
* Upper or lower respiratory tract infection (viral or bacterial) within the 2 weeks prior to Screening and Baseline Visits.
* History of clinically significant renal, hepatic, cardiovascular, metabolic, neurologic, hematologic, ophthalmologic, respiratory, gastrointestinal, cerebrovascular, or other significant medical illness or disorder which, in the judgment of the investigator, could interfere with the study or require treatment that might interfere with the study. Specific examples include but are not limited to insulin-dependent diabetes, hypertension, active hepatitis, cardiovascular disease including hypertension, or conditions that may interfere with respiratory function such as, bronchiectasis, and cystic fibrosis. Other conditions that are well controlled and stable will not prohibit participation if deemed appropriate per the investigator's judgment.
* Inability to correctly use an oral MDI or a DPI.
* Participation in this study at another investigational site. Participation in a different investigational study at any site during the same time frame of this study.
* Randomization into this study more than once.
* Direct association with either the administration of the this study or the study staff.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 583 (Actual)
Dates: Start 2012-01-25 (Actual); Primary Completion 2015-01-29 (Actual); Study Completion 2015-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amar NJ, Shekar T, Varnell TA, Mehta A, Philip G. Mometasone furoate (MF) improves lung function in pediatric asthma: A double-blind, randomized controlled dose-ranging trial of MF metered-dose inhaler. Pediatr Pulmonol. 2017 Mar;52(3):310-318. doi: 10.1002/ppul.23563. Epub 2016 Oct 14. PMID 27740721

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 583 participants were randomized; 5 participants were randomized in error and did not receive any doses of randomized study drug.
Groups:
- MF MDI 50 mcg BID: Participants receive mometasone furoate (MF) metered dose inhaler (MDI) 25 mcg x 2 inhalations (50 mcg total dose) twice daily (BID) PLUS Placebo dry powder inhaler (DPI) x 1 inhalation once daily (QD) in the evening for 12 weeks.
Period: Overall Study
Arm/Group | MF MDI 50 mcg BID | MF MDI 100 mcg BID | MF MDI 200 mcg BID | MF DPI 100 mcg QD | Placebo
Started | 120 | 113 | 108 | 125 | 112
Completed | 79 | 81 | 83 | 88 | 60
Not Completed | 41 | 32 | 25 | 37 | 52
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 1 | 1
Not completed — Adverse Event | 2 | 1 | 0 | 4 | 3
Not completed — Treatment Failure | 22 | 20 | 12 | 19 | 30
Not completed — Lack of Efficacy | 3 | 3 | 2 | 2 | 4
Not completed — Physician Decision | 3 | 0 | 0 | 0 | 1
Not completed — Noncompliance with Study Drug | 0 | 0 | 1 | 2 | 1
Not completed — Technical Problems | 1 | 0 | 2 | 4 | 1
Not completed — Protocol Violation | 9 | 5 | 6 | 5 | 10
Not completed — Excluded Medication | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of all randomized participants who received at least one dose of randomized study drug.
Groups:
- MF MDI 50 mcg BID: Participants receive MF MDI 25 mcg x 2 inhalations (50 mcg total dose) BID PLUS Placebo DPI x 1 inhalation QD in the evening for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | MF MDI 50 mcg BID | MF MDI 100 mcg BID | MF MDI 200 mcg BID | MF DPI 100 mcg QD | Placebo | Total
Number analyzed (Participants) | 120 | 113 | 108 | 125 | 112 | 578
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.7 (1.7) | 8.6 (1.9) | 8.7 (1.7) | 8.7 (1.7) | 9.0 (1.7) | 8.8 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 44 | 59 | 48 | 30 | 232
  Male | 69 | 69 | 49 | 77 | 82 | 346

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent Predicted Morning (AM) Forced Expiratory Volume in 1 Second (FEV1) - MF MDI vs. Placebo
Description: FEV1 is the amount of air, measured in liters, forcibly exhaled in 1 second. Pulmonary function tests were to be performed by participants in the morning before dosing. The percent predicted FEV1 equals the participant's observed FEV1 divided by the participant's predicted FEV1 (determined by height and race) and converted to a percentage by multiplying by 100%. The goal of the primary outcome measure was to compare the change from Baseline in AM FEV1 between the MF MDI and Placebo treatment groups. The comparison between the MF MDI 50 mcg BID vs. MF DPI 100 mcg QD treatment groups is presented in a subsequent outcome measure.
Time Frame: Baseline and Week 12
Population: The Full Analysis Set (FAS) population consisted of all participants who received ≥1 study drug dose and had a Baseline or ≥1 post-randomization value for this outcome measure. Only participants who received MF MDI or Placebo were included in this primary analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Predicted FEV1
Arm/Group | MF MDI 50 mcg BID | MF MDI 100 mcg BID | MF MDI 200 mcg BID | Placebo
Number analyzed (Participants) | 114 | 109 | 105 | 111
Percentage of Predicted FEV1 | 4.52 [2.32 to 6.72] | 6.95 [4.73 to 9.16] | 6.00 [3.74 to 8.25] | 0.66 [-1.72 to 3.03]
Statistical Analysis 1: Comparison: MF MDI 50 mcg BID vs Placebo; Change from Baseline in percent predicted FEV1 at Week 12: MF MDI 50 mcg BID vs. Placebo; Test type: Superiority or Other; p = 0.019, cLDA model — Constrained longitudinal data analysis (cLDA) model method proposed by Liang & Zeger includes terms for treatment, time in weeks, age strata (age 5-6, 7-11), treatment by time interaction & region (North America, Latin America & the European Union); Mean Difference (Net) = 3.87, 95% CI 2-sided [0.64 to 7.09]
Statistical Analysis 2: Comparison: MF MDI 100 mcg BID vs Placebo; Change from Baseline in percent predicted FEV1 at Week 12: MF MDI 100 mcg BID vs. Placebo; Test type: Superiority or Other; p < 0.001, cLDA — cLDA model method proposed by Liang & Zeger includes terms for treatment, time in weeks, age strata (age 5-6, 7-11), treatment by time interaction & region (North America, Latin America & the European Union); Mean Difference (Net) = 6.29, 95% CI 2-sided [3.05 to 9.53]
Statistical Analysis 3: Comparison: MF MDI 200 mcg BID vs Placebo; Change from Baseline in percent predicted FEV1 at Week 12: MF MDI 200 mcg BID vs. Placebo; Test type: Superiority or Other; p = 0.001, cLDA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 5.34, 95% CI 2-sided [2.07 to 8.61]

2. Secondary Outcome: Change From Baseline in AM Peak Expiratory Flow (PEF) - MF MDI vs. Placebo
Description: PEF, measured in liters per minute, is the highest flow during exhalation. Participants recorded diary entries for PEF twice daily (in the morning upon rising and in the evening at bedtime). The goal of the secondary outcome measure was to compare the change from Baseline in AM PEF between the MF MDI and Placebo treatment groups.
Time Frame: Baseline and Week 12
Population: The FAS population consisted of all participants who received ≥1 study drug dose and had a Baseline or ≥1 post-randomization value for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/minute
Arm/Group | MF MDI 50 mcg BID | MF MDI 100 mcg BID | MF MDI 200 mcg BID | Placebo | MF DPI 100 mcg QD
Number analyzed (Participants) | 118 | 112 | 108 | 111 | 123
Liters/minute | 17.83 [5.35 to 30.3] | 26.03 [13.55 to 38.51] | 16.68 [4.50 to 28.86] | -1.32 [-15.49 to 12.85] | -0.92 [-12.82 to 10.99]
Statistical Analysis 1: Comparison: MF MDI 50 mcg BID vs Placebo; Change from Baseline in AM PEF: MF MDI 50 mcg BID vs. Placebo. Only participants who received MF MDI or Placebo were included in the statistical analysis; Test type: Superiority or Other; p = 0.045, cLDA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 19.15, 95% CI 2-sided [0.43 to 37.87]
Statistical Analysis 2: Comparison: MF MDI 100 mcg BID vs Placebo; Change from Baseline in AM PEF: MF MDI 100 mcg BID vs. Placebo. Only participants who received MF MDI or Placebo were included in the statistical analysis; Test type: Superiority or Other; p = 0.004, cLDA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 27.35, 95% CI 2-sided [8.63 to 46.08]
Statistical Analysis 3: Comparison: MF MDI 200 mcg BID vs Placebo; Change from Baseline in AM PEF: MF MDI 200 mcg BID vs. Placebo. Only participants who received MF MDI or Placebo were included in the statistical analysis; Test type: Superiority or Other; p = 0.057, cLDA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 18.01, 95% CI 2-sided [-0.51 to 36.53]

3. Secondary Outcome: Change From Baseline in Paediatric Asthma Quality of Life Questionnaire With Standardised Activities (PAQLQ(S)) Total Score - MF MDI vs. Placebo
Description: The PAQLQ(S) consists of 23 questions in 3 categories: Symptoms (10 items), Activity Limitations (5 items), and Emotional Function (8 items). Responses are based on a 7-point scale (7=not bothered at all to 1=extremely bothered). PAQLQ(S) Total Scores could range from 23 to 161, with a lower score indicating a lower quality of life. The PAQLQ(S) included only participants in participating countries in which a validated translated questionnaire was available. The goal of the secondary outcome measure was to compare the change from Baseline in PAQLQ(S) between the MF MDI and Placebo treatment groups.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MF MDI 50 mcg BID | MF MDI 100 mcg BID | MF MDI 200 mcg BID | Placebo | MF DPI 100 mcg QD
Number analyzed (Participants) | 111 | 105 | 101 | 102 | 115
Score on a Scale | 0.35 [0.23 to 0.48] | 0.38 [0.25 to 0.50] | 0.44 [0.31 to 0.56] | 0.26 [0.12 to 0.39] | 0.47 [0.35 to 0.59]
Statistical Analysis 1: Comparison: MF MDI 50 mcg BID vs Placebo; Change from Baseline in PAQLQ(S) Total Score: MF MDI 50 mcg BID vs. Placebo. Only participants who received MF MDI or Placebo were included in the statistical analysis; Test type: Superiority or Other; p = 0.280, cLDA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.08 to 0.27]
Statistical Analysis 2: Comparison: MF MDI 100 mcg BID vs Placebo; Change from Baseline in PAQLQ(S) Total Score: MF MDI 100 mcg BID vs. Placebo. Only participants who received MF MDI or Placebo were included in the statistical analysis; Test type: Superiority or Other; p = 0.178, cLDA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.06 to 0.30]
Statistical Analysis 3: Comparison: MF MDI 200 mcg BID vs Placebo; Change from Baseline in PAQLQ(S) Total Score: MF MDI 200 mcg BID vs. Placebo. Only participants who received MF MDI or Placebo were included in the statistical analysis; Test type: Superiority or Other; p = 0.045, cLDA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.18, 95% CI 2-sided [0.00 to 0.36]

4. Secondary Outcome: Change From Baseline in Percent Predicted AM FEV1 - MF MDI 50 mcg BID vs. MF DPI 100 mcg QD
Description: FEV1 is the amount of air, measured in liters, forcibly exhaled in 1 second. Pulmonary function tests were to be performed by participants in the morning before dosing. The percent predicted FEV1 equals the participant's observed FEV1 divided by the participant's predicted FEV1 (determined by height and race) and converted to a percentage by multiplying by 100%. The goal of the secondary outcome measure was to compare the change from Baseline in AM FEV1 between the MF MDI 50 mcg BID and MF DPI 100 mcg QD treatment groups. The comparisons between the other MF MDI BID and Placebo treatment groups are presented in a previous outcome measure.
Time Frame: Baseline and Week 12
Population: The FAS population consisted of all participants who received ≥1 study drug dose and had a Baseline or ≥1 post-randomization value for this outcome measure. Only participants who received MF MDI 50 mcg or MF DPI were included in this secondary analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Predicted FEV1
Arm/Group | MF MDI 50 mcg BID | MF DPI 100 mcg QD
Number analyzed (Participants) | 114 | 122
Percentage of Predicted FEV1 | 4.52 [2.32 to 6.72] | 3.13 [1.01 to 5.25]
Statistical Analysis 1: Comparison: MF MDI 50 mcg BID vs MF DPI 100 mcg QD; Change from Baseline in percent predicted FEV1 at Week 12: MF MDI 50 mcg BID vs. MF DPI 100 mcg QD. Only participants who received MF MDI 50 mcg BID or MF DPI 100 mcg QD were included in the statistical analysis; Test type: Superiority or Other; p = 0.368, cLDA model — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 1.39, 95% CI 2-sided [-1.65 to 4.44]

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: The Safety population consisted of all participants who received at least one dose of randomized study drug.
Arm/Group | MF MDI 50 mcg BID | MF MDI 100 mcg BID | MF MDI 200 mcg BID | MF DPI 100 mcg QD | Placebo
Serious Adverse Events (participants affected / at risk) | 2/120 | 1/113 | 2/108 | 4/125 | 2/112
Other Adverse Events (participants affected / at risk) | 19/120 | 18/113 | 18/108 | 16/125 | 19/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF MDI 50 mcg BID (N=120) | MF MDI 100 mcg BID (N=113) | MF MDI 200 mcg BID (N=108) | MF DPI 100 mcg QD (N=125) | Placebo (N=112)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF MDI 50 mcg BID (N=120) | MF MDI 100 mcg BID (N=113) | MF MDI 200 mcg BID (N=108) | MF DPI 100 mcg QD (N=125) | Placebo (N=112)
Nasopharyngitis (Infections and infestations) | 8 (9) | 5 (6) | 7 (9) | 8 (8) | 8 (9)
Accidental overdose (Injury, poisoning and procedural complications) | 13 (18) | 13 (19) | 12 (19) | 10 (14) | 13 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.